CLINICAL TRIAL: NCT07167511
Title: Efficacy and Safety of Bismuth-containing Quadruple Therapy for First Line Helicobacter Pylori Eradication: A Multicenter Retrospective Study
Brief Title: Bismuth-containing Quadruple Therapy for Helicobacter Pylori Eradication
Acronym: RETRO-HP
Status: Completed | Type: Observational
Sponsor: Yueyue Li (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Zaozhuang Municipal Hospital (Other); Shandong University of Traditional Chinese Medicine (Other); Qihe County People's Hospital (Unknown); Taierzhuang District People's Hospital (Other); University Town Hospital, Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Unknown); Dezhou Hospital Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor-Investigator, Yueyue Li, Associate Professor, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Other Study IDs: 202508
Record Dates: First submitted 2025-08-25; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; quadruple therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- vonoprazan-based quadruple therapies
  Interventions: Other: This study is a retrospective study, and all data have been collected in advance with no active intervention required.
- tegoprazan-based quadruple therapies
  Interventions: Other: This study is a retrospective study, and all data have been collected in advance with no active intervention required.

INTERVENTIONS:
Other: This study is a retrospective study, and all data have been collected in advance with no active intervention required. — This study is a retrospective study, and all data have been collected in advance with no active intervention required.

SUMMARY:
Bismuth-containing quadruple therapy was recommended as a first-line treatment for Helicobacter pylori infection. This study aimed to compare real-world outcomes of various bismuth-containging quadruple regimens and identify factors influencing treatment failure. A multicenter retrospective analysis was conducted and study outcomes included eradication rates and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-70 years, regardless of gender;
* absent history of receiving H. pylori eradication therapy;
* diagnosed with H. pylori infection through at least one of the following methods: rapid urease test, ¹³C/¹⁴C-urea breath test, or histopathological examination.

Exclusion Criteria:

* patients with incomplete medical records, including missing treatment details, absence of post-treatment follow-up test results, or failure to complete essential follow-up assessments;
* patients who received treatment regimens that did not comply with the quadruple regimens specified in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) patients aged 18-70 years, regardless of gender; (2) absent history of receiving H. pylori eradication therapy; (3) diagnosed with H. pylori infection through at least one of the following methods: rapid urease test, ¹³C/¹⁴C-urea breath test, or histopathological examination.
Sampling Method: Non-Probability Sample
Enrollment: 1730 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Eradication rate | 6 weeks after treatment completion
  Comparison of eradication rates among quadruple therapies for Helicobacter pylori

SECONDARY OUTCOMES:
Adverse events | Immediately after treatment completion

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China